CLINICAL TRIAL: NCT06567041
Title: Investigation of the Safety, Tolerability, Pharmacokinetics and Efficacy of Subcutaneous Weekly Doses of NNC0519-0130 in Participants With Obesity and in Participants With Type 2 Diabetes With Either Overweight or Obesity
Brief Title: A Research Study of How Safe a New Medicine Called NNC0519 0130 is and to Test Its Effect in People Living With Excess Body Weight With or Without Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9541-8116; U1111-1305-5164 (Other: Universal Trial Number); 2024-512719-28 (Other: EU CT Number)
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0519-0130 (Experimental): Participants will receive NNC0519-0130 once weekly (QW) subcutaneously(s.c.).
  Interventions: Drug: NNC0519-0130
- Placebo (Placebo Comparator): Participants will receive once weekly s.c. volume-matched placebo to NNC0519-0130.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0519-0130 — NNC0519-0130 will be administered subcutaneously.
  Arms: NNC0519-0130
Drug: Placebo — Placebo will be administered subcutaneously.
  Arms: Placebo

SUMMARY:
A new study medicine called NNC0519-0130 to improve treatment options for people living with excess body weight, with or without type 2 diabetes. The purpose of the study is to investigate potential side effects and blood levels of NNC0519-0130, as well as changes in body weight, blood sugar levels, and heart activity. The study consists of two groups, with participants receiving either the study medicine (NNC0519-0130) or a placebo. Which treatment participants get is decided by chance and they can only participate in one group. Participants will be given the study medicine once weekly, and it should be taken on the same day each week. The treatment duration depends on the group participants are enrolled in, with the study lasting for 37 weeks for Group 1 and 34 weeks for Group 2.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female of non-childbearing potential.
* Age 18-55 years (both inclusive) at the time of signing the informed consent.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Participants with obesity only:

* Body mass index between 30.0 kilogram per meter square (kg/m^2) and 39.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.

Participants with type 2 diabetes with either overweight or obesity:

* Body mass index between 27.0 kg/m^2 and 39.9kg/m^2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Diagnosed with type 2 diabetes mellitus greater than or equal to (≥) 180 days before screening.
* Glycated haemoglobin (HbA1c) in the range of 6.5 percentage (%) (inclusive) and 9.5% (inclusive).

Exclusion Criteria:

* Any condition, except T2D and hypertension, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological conditions (except diabetes mellitus and hypertension).
* Presence or history of cardiovascular disease including stable and unstable angina pectoris, myocardial infarction, transient ischaemic attack, stroke, cardiac decompensation, clinically significant arrhythmias or clinically significant conduction disorders.
* Participant is breastfeeding.

Participants with obesity only:

* HbA1c ≥ 6.5 % (48 millimoles per mol [mmol/mol]) at screening.

Participants with type 2 diabetes with either overweight or obesity:

* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Recurrent severe hypoglycaemia within the last year as judged by the investigator.
* Known hypoglycaemic unawareness as indicated by the investigator according to Clarke's questionnaire question 8.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | From time of first dosing (day 1) until completion of the end of study visit (day 274/253)
  Measured in number of events.

SECONDARY OUTCOMES:
Change in 12-lead electrocardiogram, Individual-specific heart rate corrected QT interval (QTcI) | From baseline (day - 1) until completion of the end of study visit (day 274/253)
  Measured in milliseconds (ms).
Change in 12-lead electrocardiogram, Fridericia heart rate corrected QT interval (QTcF) | From baseline (day - 1) until completion of the end of study visit (day 274/253)
  Measured in ms.
Area under the NNC0519-0130 plasma concentration-time curve in steady state | From pre-dose until 7 days post-dose, for third and last doses in the maintenance period
  Measured in hours*nanomoles per liter (h*nmol/L).
Maximum plasma concentration of NNC0519-0130 in steady state | From pre-dose until 7 days post-dose, for third and last doses in the maintenance period
  Measured in nanomoles per liter (nmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Parexel International GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com